CLINICAL TRIAL: NCT00888355
Title: A Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Investigate the Antihypertensive Efficacy and Safety of Losartan Given Once or Twice Daily in Patients With Mild to Moderate Hypertension
Brief Title: MK0954 Versus Placebo for Treatment of Mild to Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009_582; MK0954-065
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2009-06-24 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo
- 2 (Experimental): Losartan 50 q.a.m.
  Interventions: Drug: losartan potassium
- 3 (Experimental): Losartan 25 b.i.d.
  Interventions: Drug: losartan potassium
- 4 (Experimental): Losartan 25 q.a.m.
  Interventions: Drug: losartan potassium

INTERVENTIONS:
Drug: losartan potassium — losartan tablet (MK0954) 25 or 50 mg q.a.m. or 25 mg b.i.d., for 12 weeks
  Other Names: MK0954
  Arms: 2; 3; 4
Drug: Comparator: placebo — placebo to losartan tablet q.a.m. , for 12 weeks
  Arms: 1

SUMMARY:
The study had a 4 week single blind placebo period followed by 12 weeks of double blind treatment. Patients were randomized to one of four treatment arms to evaluate the antihypertensive efficacy of Losartan.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with mild to moderate hypertension
* Patient has no treatment or active medical problem, other than hypertension that might affect the patients blood pressure

Exclusion Criteria:

* Pregnant of lactating female patients
* Secondary hypertension or history of malignant hypertension
* Sitting systolic blood pressure > 210 mmHg
* History of stroke
* History of myocardial infarction with in the past year
* Current of prior history of heart failure
* Known hypersensitivity to losartan
* Obesity
* Patients known to be HIV positive or known to be positive for Hepatitis B
* Absence of one kidney
* Patient is abusing or previously abused alcohol or drugs with in past two years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 1992-05; Primary Completion 1993-01 (Actual); Study Completion 1993-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 37 sites in the United States. Prime Therapy Period: May, 1992 to January1993
Pre-assignment Details: Patients could be randomized if sitting diastolic blood pressure (SiDBP) after 2 and 4 weeks of placebo washout was 95-115 mm Hg and the difference between measurements at the 2 visits did not differ by >7 mm Hg.
Groups:
- Placebo: Losartan placebo orally once daily for 12 weeks
- Losartan 25 mg q.d.: Losartan 25 mg orally once daily (q.d.) for 12 weeks
- Losartan 50 mg q.d.: Losartan 50 mg orally once daily (q.d.) for 12 weeks
- Losartan 25 mg (b.i.d.): Losartan 25 mg orally twice daily (b.i.d.) for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Started | 108 | 108 | 106 | 106
Completed | 86 | 99 | 94 | 96
Not Completed | 22 | 9 | 12 | 10
Not completed — Adverse Event | 10 | 0 | 3 | 3
Not completed — Lack of Efficacy | 9 | 2 | 5 | 2
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0
Not completed — Protocol Violation | 3 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.) | Total
Number analyzed (Participants) | 108 | 108 | 106 | 106 | 428
Age Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.6) | 53.0 (10.7) | 54.0 (10.1) | 52.4 (10.1) | 53.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 36 | 36 | 151
  Male | 70 | 67 | 70 | 70 | 277
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 84 | 79 | 82 | 89 | 334
  Oriental | 1 | 2 | 2 | 2 | 7
  Latin American | 0 | 1 | 0 | 0 | 1
  Black | 21 | 22 | 17 | 10 | 70
  Hispanic | 2 | 4 | 5 | 4 | 15
  Vietnamese | 0 | 0 | 0 | 1 | 1
Sitting Diastolic Blood Pressure (SiDBP) [Mean (Standard Deviation); unit: mm Hg] | 101.5 (5.1) | 101.8 (5.5) | 102.4 (6.4) | 102.0 (5.3) | 101.9 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Mean change from baseline in trough (24 hours after the last morning dose and 12 hours after the last PM dose) SiDBP at Week 12
Time Frame: At baseline, and at 12 weeks (24 hours after last morning dose and 12 hours after last PM dose)
Population: The primary analysis employed an "all patients treated" approach that included patients with at least one treatment period measurement. The last measurements of withdrawn patients were carried forward to subsequent timepoints. Missing data were estimated by carrying forward data from the last visit (excluding baseline) at which it was available.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 102 | 105 | 101 | 101
mm Hg | -2.0 (8.4) | -5.8 (6.7) | -6.3 (7.4) | -8.0 (7.9)

2. Secondary Outcome: Mean Change From Baseline in Trough Sitting Systolic Blood Pressure (SiSBP) as Week 12
Description: Mean change from baseline in trough (24 hours after the last morning dose and 12 hours after the last PM dose) SiSBP at Week 12
Time Frame: At baseline, and at 12 weeks (24 hours after last morning dose and 12 hours after last PM dose)
Population: An "all patients treated" approach was employed that included patients with at least one treatment period measurement. The last measurements of withdrawn patients were carried forward to subsequent timepoints. Missing data were estimated by carrying forward data from the last visit (excluding baseline) at which it was available.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 102 | 105 | 101 | 101
mm Hg | -0.2 (15.1) | -7.2 (13.9) | -7.6 (12.6) | -8.8 (13.0)

3. Secondary Outcome: Mean Change From Baseline in Peak Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Mean change from baseline in peak (6 hours after the last morning dose) SiDBP at Week 12
Time Frame: At baseline and at 12 weeks (6 hours after last morning dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 92 | 95 | 94 | 94
mm Hg | -3.0 (9.7) | -7.7 (8.5) | -8.7 (8.1) | -9.9 (9.5)

4. Secondary Outcome: Categories of Antihypertensive Response in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Patients with trough SiDBP <90 mm Hg were in Category I, ≥90 but decreased at least 10 mm Hg were in Category II, and ≥90 and decreased less than 10 mm Hg or increased were in Category III.
Time Frame: 24 hours after last morning dose and 12 hours after last PM dose at 12 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 102 | 105 | 101 | 101
Participants
  Category I | 12 | 23 | 26 | 33
  Category II | 10 | 14 | 14 | 15
  Category III | 80 | 68 | 61 | 53

5. Other Pre Specified Outcome: Number of Patients With Clinical Adverse Experiences (CAEs)
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 12 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 108 | 108 | 106 | 106
Participants
  With CAEs | 63 | 59 | 59 | 60
  Without CAEs | 45 | 49 | 47 | 46

6. Other Pre Specified Outcome: Number of Patients With Serious CAEs
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 12 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 108 | 108 | 106 | 106
Participants
  With Serious CAEs | 4 | 1 | 1 | 3
  Without Serious CAEs | 104 | 107 | 105 | 103

7. Other Pre Specified Outcome: Number of Patients With Drug-related CAEs
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs during the 12-week treatment period
Time Frame: 12 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 108 | 108 | 106 | 106
Participants
  With drug-related CAEs | 20 | 12 | 21 | 16
  Without drug-related CAEs | 88 | 96 | 85 | 90

8. Other Pre Specified Outcome: Number of Patients Discontinued Due to CAEs
Description: Patients discontinued due to CAEs during the 12-week treatment period
Time Frame: 12 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 108 | 108 | 106 | 106
Participants
  Discontinued due to CAEs | 10 | 0 | 1 | 3
  Not discontinued due to CAEs | 98 | 108 | 105 | 103

9. Other Pre Specified Outcome: Number of Patients Who Died
Description: Patients who died during the 12-week treatment period
Time Frame: 12 weeks
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 108 | 108 | 106 | 106
Participants
  Who Died | 2 | 0 | 0 | 1
  Alive | 106 | 108 | 106 | 105

10. Other Pre Specified Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs)
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 12 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 104 | 105 | 103 | 104
Participants
  With LAEs | 7 | 7 | 7 | 4
  Without LAEs | 97 | 98 | 96 | 100

11. Other Pre Specified Outcome: Number of Patients With Serious LAEs
Description: Serious LAEs are any LAEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 12 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 104 | 105 | 103 | 104
Participants
  With serious LAEs | 0 | 0 | 0 | 0
  Without serious LAEs | 104 | 105 | 103 | 104

12. Other Pre Specified Outcome: Number of Patients With Drug-related LAEs
Description: Patients with drug-related LAEs during the 12-week treatment period
Time Frame: 12 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 104 | 105 | 103 | 104
Participants
  With drug-related LAEs | 4 | 5 | 4 | 0
  Without drug-related LAEs | 100 | 100 | 99 | 104

13. Other Pre Specified Outcome: Number of Patients Discontinued Due to LAEs
Description: Patients discontinued due to LAEs during the 12-week treatment period
Time Frame: 12 weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 25 mg q.d. | Losartan 50 mg q.d. | Losartan 25 mg (b.i.d.)
Number analyzed (Participants) | 104 | 105 | 103 | 104
Participants
  Discontinued due to LAEs | 0 | 0 | 2 | 0
  Not discontinued due to LAEs | 104 | 105 | 101 | 104

LIMITATIONS AND CAVEATS:
Note that deaths are not entered under "drop reasons" in the participant flow panel because the patients who died are already counted as dropped due to adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes